CLINICAL TRIAL: NCT03994627
Title: An Open-Label, Multi-Center Patient Access Program of Olaratumab for the Treatment of Soft Tissue Sarcoma
Brief Title: Olaratumab (LY3012207) Patient Access for Soft Tissue Sarcoma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 17468; I5B-MC-Y001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaratumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Olaratumab — Administered intravenously (IV)
  Other Names: LY3012207

SUMMARY:
The purpose of this study is to continue to provide olaratumab to eligible patients who are currently receiving olaratumab commercially for the treatment of soft tissue sarcoma (STS).

ELIGIBILITY:
Inclusion Criteria:

* Are currently receiving olaratumab and who, in consultation with their treating physician, want to continue their course of therapy.
* Have metastatic or locally advanced unresectable soft tissue sarcoma not amenable to curative treatment with surgery or radiotherapy.
* Have given written informed consent.
* Have an absolute neutrophil count (ANC) ≥1,000/microliter.
* Females of childbearing potential and males must agree to use highly effective contraceptive precautions during treatment with olaratumab and up to 3 months following the last dose of olaratumab. A highly effective method of birth control is defined as one that results in a low failure rate (that is, <1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomized partner.

Exclusion Criteria:

* Breastfeeding (patients who discontinue breastfeeding would be considered eligible).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (89):
- United States (55):
  - Ironwood Cancer & Research Centers, Glendale, Arizona
  - Marin Specialty Care, Inc, Greenbrae, California
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Kaiser Permanente Moreno Valley, Moreno Valley, California
  - University of Colorado Health Hospital, Aurora, Colorado
  - UCHealth Cancer Center, Fort Collins, Colorado
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Ocala Oncology, P.A., Ocala, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Orlando Health UF Health Cancer Center, Orlando, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Oncology-Hematology Associates of West Broward, Tamarac, Florida
  - Northside Hospital, Athens, Georgia
  - Tift Regional Health System Anita Stewart Oncology Center, Tifton, Georgia
  - Beacon Cancer Care, Coeur d'Alene, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Alton Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - SKCCC at Johns Hopkins, Baltimore, Maryland
  - Baltimore Washington Health Services, Glen Burnie, Maryland
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - St. Luke's Hospital of Duluth, Duluth, Minnesota
  - Masonic Cancer Center, University, Minneapolis, Minnesota
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - University of Mississippi School of Medicine, Jackson, Mississippi
  - County Oncologist, Inc., St Louis, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Regional Cancer Care Associates, LLC, East Brunswick, New Jersey
  - Hudson Valley Cancer Center, Fishkill, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - East Carolina School of Medicine, Greenville, North Carolina
  - Aultman Medical Group Hematology & Oncology, Canton, Ohio
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The James Cancer Hospital, Columbus, Ohio
  - UPMC Hillman Cancer Center, Greenville, Pennsylvania
  - Steward Sharon Regional Cancer Center, Hermitage, Pennsylvania
  - UPMC Hillman Cancer Center, New Castle, Pennsylvania
  - Abramson Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - The West Clinic, Germantown, Tennessee
  - Tennessee Oncology PLLC, Hixson, Tennessee
  - UVAHS Emily Couric Clin Cancer Ctr, Charlottesville, Virginia
  - Kaiser Permanente of WA, Olympia, Washington
  - Harrison HealthPartners Hematology, Poulsbo, Washington
  - Seattle Integrative Cancer Center, Renton, Washington
  - Mon Health Medical Center, Morgantown, West Virginia
  - SSM Health Cancer Care Center, Madison, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin
- Austria (2):
  - Ordensklinikum Linz GmbH Elisabethinen, Linz, Upper Austria
  - Kepler Universitätsklinikum GmbH, Med Campus III, Linz, Upper Austria
- Brazil (2):
  - CLION - Clínica de Oncologia, Salvador, Estado de Bahia
  - Instituto Londrina de Radioterapia, Londrina, Paraná
- Canada (2):
  - CHUM, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Hungary (2):
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Jósa András Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - National Institute of Oncology, Budapest
- Healthcare Global Enterprises Limited (HCG), Bangalore, Karnataka, India
- Italy (3):
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - IRCCS - AOU di Bologna, Bologna
  - Ospedale Santa Chiara di Trento, Trento
- South Korea (5):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon
  - Inha University Hospital, Incheon, Incheon-gwangyeoksi [Incheon]
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Pusan National University Hospital, Busan, Pusan-Kwangyǒkshi
  - Wonkwang University Hospital, Iksan-si, Jeonlabuk-do
- Spain (12):
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, La Laguna
  - Hospital De Navarra, Pamplona, Navarre
  - Clínica Mompia, Cantabria, Santa Cruz de Bezana
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Cl. Universitaria Navarra, Madrid
  - Centro Oncológico MD Anderson, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Gerencia de Asistencia Sanitaria de Segovia_Hospital General de Segovia, Segovia
  - Hospital Universitario Virgen Del Rocio, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario La Fe de Valencia, Valencia
- China Medical University Hospital, Taichung, Taiwan
- United Kingdom (4):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Ninewells Hospital, Dundee, Scotland
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge